CLINICAL TRIAL: NCT01032616
Title: Determination of the Difference in Uptake and Utilization of Two Amino Acids by the Splanchnic Bed
Brief Title: Uptake and Utilization of Amino Acids by Splanchnic Bed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Karen Chapman, Clinical Research Nurse Specialist, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0019880597 (Part b)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Healthy Males
Keywords: splanchnic bed; theronine and lysine metabolism uptake; isotopes; metabolism of two indispensable amino acids, threonine and lysine, by the splanchnic bed by Healthy Males

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Period 1 (Experimental): AA given by parenteral and enteral routes with tracer 1-13C phenylalanine given to observe differences
  Interventions: Other: Threonine Experimental: Study Period 1
- Study Period 2 (Experimental): AA given by parenteral and enteral routes with tracer 1-13C phenylalanine given to observe differences
  Interventions: Other: Lysine Experimental: Study Period 2

INTERVENTIONS:
Other: Threonine Experimental: Study Period 1 — Enteral and parenteral infusion of threonine isotope
  Other Names: Tracer Isotope - L-[1-13C]threonine
  Arms: Study Period 1
Other: Lysine Experimental: Study Period 2 — Both intravenous (iv) and intragastric (ig) Lysine isotopes.
  Other Names: Tracer isotope - L-[1-13C]lysine
  Arms: Study Period 2

SUMMARY:
Splanchnic uptake and metabolism contributes significantly to the differences in flux seen between the intravenous and intragastric ingestion of certain indispensable amino acids.

This is the third in a series of studies designed to increase the investigators knowledge of the metabolism of two indispensable amino acids, threonine and lysine, by the splanchnic bed. In the initial two studies the investigators established the neonatal parenteral requirement of threonine and lysine. In the current study, the investigators will be examining the differences in uptake and metabolism of threonine and lysine across the splanchnic bed.

DETAILED DESCRIPTION:
We propose that we will see a smaller amount of enterally fed isotopes reach the plasma as compared to the amount in plasma from the parenterally delivered isotopes. We also believe that the amount of enterally delivered threonine isotope that reaches the plasma will be significantly less than the amount of enterally fed lysine isotope.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Males

Exclusion Criteria:

* History of inborn error of metabolism
* Presence of a chronic disease
* Have unusual dietary practices
* Has recently lost weight
* Receiving pharmacological therapy or hormonal treatment

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Breath VCO2 | -30min, -20min, -10min, +2.5hrs, +3 hrs, +3.5hrs, +4hrs,+4.5hrs, +5hrs
Blood CO2 | -30min, -20min, -10min, +2.5hrs, +3 hrs, +3.5hrs, +4hrs,+4.5hrs, +5hrs

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pencharz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada